CLINICAL TRIAL: NCT02030886
Title: A Single-center, Open Label, Prospective Study Assessing the 24-hour IOP Patterns Using SENSIMED Triggerfish® in Ocular Hypertensive Patients Newly Converted to Glaucomatous Disease Versus Stable Ocular Hypertensive Patients
Brief Title: IOP Patterns in Ocular Hypertensive Patients Newly Converted to Glaucoma vs Stable Ocular Hypertensive Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Sensimed AG (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TF-1302
Record Dates: First submitted 2013-12-30; First posted 2014-01-09 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ocular hypertension subjects (Other): All subjects will be monitored by Sensimed Triggerfish (TF) for 24 hours.
  Interventions: Device: Sensimed Triggersfish® (TF)

INTERVENTIONS:
Device: Sensimed Triggersfish® (TF) — All subjects will be monitored by Sensimed Triggerfish (TF) for 24 hours.

SUMMARY:
The purpose of the study is to assess the relationship between IOP pattern as recorded over 24 hours by using Triggerfish and quantified by acrophase scored dichotomously, and conversion to glaucoma in OHT patients (conversion status). Elevation of IOP above normal range is called "ocular hypertension" (OHT). In a previous study, it has been shown that OHT patients who progress to glaucoma (converters) have at baseline and prior to any conversion, IOP patterns that more closely resemble those of established early primary open-angle glaucoma (POAG) patients, while stable OHT patients (non-converters) have IOP patterns closer to those of healthy control subjects. The study has been planned to recruit at least 48 eligible patients (24 converters and 24 non-converters).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OHT (IOP >21 mmHg on 2 consecutive visits) in the study eye
* No IOP-lowering drug treatment in the study eye; otherwise, a 4-week wash-out period prior to study day 0 (SD0) and throughout the study
* Aged ≥ 18 years, of either sex
* Not more than 6 diopters spherical equivalent in the study eye
* Having given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Narrow iridocorneal angle or any other concomitant ocular conditions (except cataract) in the study eye
* History of ocular surgery on the study eye (except cataract extraction)
* History of laser treatment on the study eye
* Corneal or conjunctival abnormality in the study eye, precluding contact lens adaptation
* Severe dry eye syndrome
* Subjects with irregular sleep schedules
* Subjects who are current smokers
* Subjects with allergy to corneal anesthetic
* Subjects with contraindications for silicone contact lens wear
* Subjects not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks
* Any other contra-indication listed in the TF user manual

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Liu, MD, Principal Investigator — Yale University
Locations (1):
- Yale Medical School, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ocular Hypertension Non Converters: Stable ocular hypertension patients monitored by Triggerfish (TF) for 24 hours.
- Ocular Hypertension Converters: Ocular hypertension patients who progressed to glaucoma monitored by TF for 24 hours
Period: Overall Study
Arm/Group | Ocular Hypertension Non Converters | Ocular Hypertension Converters
Started | 14 | 6
Completed | 14 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Stable ocular hypertension patients and ocular hypertension patients who progressed to glaucoma, both monitored by TF for 24 hours.
Groups:
- Ocular Hypertension Non Converters: Stable ocular hypertension patients monitored by TF for 24 hours.
- Total: Total of all reporting groups
Arm/Group | Ocular Hypertension Non Converters | Ocular Hypertension Converters | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.9) | 59.3 (6.7) | 58.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between Intraocular Pressure (IOP) Pattern as Recorded by TF, and Quantified by Acrophase Scored Dichotomously, and Conversion to Glaucoma in Ocular Hypertension (OHT) Patients (Conversion Status)
Description: For each subject, TF acrophase (ie. time when peak occured) was scored dichotomously (before and after 7 am) and compared between OHT converters and non converters patients.
  One subject was removed from the analysis because of invalid TF output.
Time Frame: 24 hours
Population: Stable ocular hypertension patients and ocular hypertension patients who progressed to glaucoma both monitored by TF for 24 hours. One subject was removed from the analysis because of invalid TF output.
Measure: Number; unit: percentage of participants
Arm/Group | Ocular Hypertension Non Converters | Ocular Hypertension Converters
Number analyzed (Participants) | 13 | 6
percentage of participants
  Before 7 am | 92.3 | 66.7
  After 7 am | 7.7 | 33.3

2. Secondary Outcome: Acrophase Scored Continuously (i.e. Actual Time of TF Peak Occurrence)
Description: Mean TF acrophase (ie. actual time when peak occured) was compared between OHT converters and non converters.
  One subject was removed from the analysis because of invalid TF output.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Ocular Hypertension Non Converters | Ocular Hypertension Converters
Number analyzed (Participants) | 13 | 6
hour | 5.35 (2.01) | 6.30 (3.55)

3. Secondary Outcome: Amplitude of Best-fitting Cosine Curve to 24-hour TF Measurements
Description: This represents an estimate of the magnitude of 24-hour IOP-related variation. One subject was removed from the analysis because of invalid TF output.
Time Frame: 24 hours
Population: Stable ocular hypertension patients and ocular hypertension patients who progressed to glaucoma, both monitored by TF for 24 hours.
  One subject was removed from the analysis because of invalid TF output.
Measure: Mean (Standard Deviation); unit: mVEq
Groups:
- Ocular Hypertension Non Converters: Stable ocular hypertension patients
- Ocular Hypertension Converters: Ocular hypertension patients who progressed to glaucoma
Arm/Group | Ocular Hypertension Non Converters | Ocular Hypertension Converters
Number analyzed (Participants) | 13 | 6
mVEq | 126.9 (52.6) | 128.0 (49.5)

ADVERSE EVENTS:
Time Frame: Within the 24h recording
Groups:
- Ocular Hypertension Non Converters: Stable ocular hypertension patients monitored by TF for 24 hours. One subject was removed from the analysis because of invalid TF output.
Arm/Group | Ocular Hypertension Non Converters | Ocular Hypertension Converters
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6
Other Adverse Events (participants affected / at risk) | 1/13 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocular Hypertension Non Converters (N=13) | Ocular Hypertension Converters (N=6)
Upper lid swelling (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No